CLINICAL TRIAL: NCT05272020
Title: PRognosis of Outcome and Recuperation of Cardiac Hemodynamic Function After Aortic Valve REplacement in Aortic Valve Stenosis
Brief Title: Outcome, Recuperation and Hemodynamics in Aortic Stenosis
Acronym: PROCARE-AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Sarah Hoedemakers, Sarah Hoedemakers, Jessa Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: f/2020/173
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVI (Other): Cardiopulmonary exercise testing, 6 minute walking test, QOL assessment
  Interventions: Diagnostic Test: CPET, 6MWT, QOL assessment
- AVR (Other): Cardiopulmonary exercise testing, 6 minute walking test, QOL assessment, Myocardial + aortic valve biopsy
  Interventions: Diagnostic Test: CPET, 6MWT, QOL assessment

INTERVENTIONS:
Diagnostic Test: CPET, 6MWT, QOL assessment — Preoperative and postoperative (6 months + 18 months) assessment

SUMMARY:
Indication for aortic valve replacement (AVR) in aortic stenosis (AS) is currently based on the classical triad of clinical AS symptoms, estimation of AS severity, and cardiac repercussion at rest. However, presence of symptoms in elderly is often subjective and underreported, and cardiac function analysis at rest underestimates the true impact of the chronic afterload increase. This complicates the diagnosis and hampers timely aortic valve replacement therapy with an impact on prognosis and cardiac function recovery. Exercise imaging in AS may reveal underlying cardiac repercussion and symptoms at an earlier stage and therefore impact prognosis and cardiac function recovery after AVR. Therefore the principal objective of this study is to reveal the factors that determine clinical outcome and hemodynamic function recovery after AVR in AS.

ELIGIBILITY:
Inclusion Criteria:

* Every patient above 18 years of age with an echocardiographic established moderate to severe AS
* A guideline indication for aortic valve replacement therapy

Exclusion Criteria:

* Unable to perform exercise testing
* Previous aortic valve intervention
* More than moderate other valvular disease
* Patients refusing participation or unwilling to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Outcome defined by the occurrence of a major cardiac event | 18 months
  either
  1. Death of cardiovascular origin, or
  2. Hospitalization for heart failure, or
  3. Deterioration of hemodynamic function during an 18 month follow-up period after AVR.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Herbots, MD PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Ziekenhuis, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No